CLINICAL TRIAL: NCT02441127
Title: Diode Laser For Harvesting Subepithelial Connective Tissue Graft in The Treatment of Gingival Recession Defects: A Novel Approach to Limit Morbidity
Brief Title: Diode Laser for Harvesting Gingival Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Onur Ozcelik, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CukurovaU4
Record Dates: First submitted 2015-04-29; First posted 2015-05-12 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Gingival Recession
Keywords: free gingival graft; diode laser; donor site; mucogingival surgery
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diode laser group (Experimental): In the test sites, an aluminum, gallium, and arsenide diode laser (wavelength 810 nm and power of 1W) was applied in continuous mode.
  Interventions: Device: diode laser group
- Scalpel control group (Active Comparator): The surgical technique used in the control group was a FGG harvested by two horizontal and two vertical incisions by scalpel defining the area to be harvested .
  Interventions: Procedure: scalpel control group

INTERVENTIONS:
Device: diode laser group — the laser tip was used to remove all visible epithelium in the outer side of the defined graft area. The treatment was performed from the coronal to the apical aspect in parallel paths, and care was taken to avoid any laser contact to the palatal bone and periosteum by aiming the laser beam at a 450 angle to the palatal soft-tissue. The resultant layer on the surface was totally removed with knife and moist gauze. Then, the graft was harvested from the de-epithelized area with a 15c blade.
  Arms: Diode laser group
Procedure: scalpel control group — In the control group tissue was obtained by two horizontal and two vertical incisions defining the area to be harvested. The blade was oriented perpendicular to the bone along the coronal horizontal incision and once an adequate soft tissue thickness was obtained; it was rotated in order to be parallel to the superficial surface. The thickness of the graft was maintained uniform while proceeding apically with the blade until the FGG was harvested. The palatal wound was protected with equine-derived collagen maintained by compressive sling 5-0 sutures
  Arms: Scalpel control group

SUMMARY:
Aims: The aim of present randomized controlled clinical study was to evaluate whether the additional use of diode laser would facilitate the donor surgery, improve the palatal wound healing and reduce post-operative morbidity after the coronally advanced flap (CAF) with connective tissue (CTG) grafts.

Methods: Fifty-two patients with isolated recessions were treated. The CTG resulted from the de-epithelialization of a free gingival graft (FGG) with blade (control group) or diode laser (DL) (test group). The DL was used to de-epithelialize the outer part of the FGG and photo-biostimulate the palatal wound area. Post-operative morbidity was evaluated by using Oral health related Quality of life (QoL), smile related QoL and visual analogue scale-discomfort (VAS). Root coverage outcomes were also evaluated 6 months after operation.

DETAILED DESCRIPTION:
The procedure of connective tissue harvesting from the palate is often characterized by the challenge of obtaining the largest volume of tissue possible on one side while minimizing post-operative pain and reducing the risk of complications on the other.The present clinical study evaluated whether the additional use of diode laser would facilitate the donor surgery, improve the palatal wound healing and reduce post-operative morbidity after the bilaminar periodontal plastic surgery procedure for the treatment of isolated single gingival recession defects with no loss of interdental clinical attachment.

In the test sites, an aluminum, gallium, and arsenide diode laser (wavelength 810 nm and power of 1W) was applied in continuous mode. In the control group,a free (epithelialized) gingival graft was harvested by two horizontal and two vertical incisions defining the area. The post operative course of the patients were evaluated by visual analogical scale and the oral health impact profile

ELIGIBILITY:
Inclusion Criteria:

* Presence of identifiable buccal cemento-enamel junction;
* Presence of a step ≤ 1mm at the cemento-enamel junction level
* No contraindications for periodontal surgery and no periodontal surgery on the involved sites
* Full-mouth plaque score of <10%; full-mouth bleeding score of <15%
* No occlusal interferences.

Exclusion Criteria:

* History of periodontitis or abscess formation
* Presence of systemic disease
* Smokers
* Pregnant patients.

Ages: 21 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-10; Primary Completion 2014-04 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Oral health related quality of life | 6 months

SECONDARY OUTCOMES:
Complete root coverage | 6 months
Smile related quality of life | 6 months
Post-operative Discomfort on the Visual Analog scale | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Onur Ozcelik, PhD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Turkey (Türkiye)